CLINICAL TRIAL: NCT07233421
Title: Frequency of Hypoglycemia in Children With Beta-blocker Treated Long QT-syndrome
Acronym: LQThypo
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Foundation for Paediatric Research, Finland (Other)
Responsible Party: Principal Investigator, Elina Hakonen, MD PhD Pediatrician, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUS/2446/2024
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Long QT Syndrome; Hypoglycemia
Keywords: propranolol; beta blocker; hypoglycemia; long qt syndrome
MeSH Terms: conditions — Long QT Syndrome; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long QT-syndrome patients (Other): Children (aged 0-6 years) with genetically verified LQT1 or LQT2
  Interventions: Device: Continuous Glucose Monitoring
- Controls (Other): 0-6 year old healthy siblings of long QT-syndrome patients
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — All participants will have the continuous glucose monitoring device Dexcom G7 placed. The Dexcom G7 Glucose Monitoring System reports continuous interstitial blood glucose concentrations every 5 minutes and alerts for low glucose (<3.1 mmol/l). Sensor low alarms are verified by finger prick tests. A single sensor is used up to 10 days and the sensoring is performed twice in each participant.

SUMMARY:
The goal of this observational study is to investigate the frequency and characteristics of hypoglycemic episodes in children with long QT syndrome (LQTS) and beta-blocker treatment, specifically those receiving propranolol, compared to healthy controls. The study focuses on children under seven years with genetically confirmed LQTS and beta-blocker therapy, as well as healthy siblings as controls.

The main questions it aims to answer are:

* Does hypoglycemic episodes occur in children with LQTS who are treated with propranolol?
* Are there asymptomatic episodes of low blood glucose that could affect well-being and neurological development?
* Are there individual differences in susceptibility to hypoglycemia, and do genetic factors explain these differences?
* What is the incidence of hypoglycemia leading to emergency visits or hospitalizations among LQTS patients compared to healthy controls?

Researchers will compare children with LQTS on propranolol to healthy siblings to see if the frequency and severity of hypoglycemia differs between groups.

Participants will:

Have a Dexcom G7 continuous glucose monitor installed to record glucose profiles for ten days, both during an healthy episode and during an infection (when risk for hypoglycemia is increased).

If differences in susceptibility to hypoglycemia are observed, genetic data from the Helsinki biopank will be analyzed to explore potential genetic factors underlying these differences. Visits to emergency clinic and hospitalizations due to hypoglycemia will be retrospectively reviewed for all LQTS patients under 16 years old and compared to healthy controls.

Additional Details:

The study is conducted at Helsinki University Hospital (HUH) Children and Adolescents and the New Children's Hospital clinical research unit. The study aims to recruit 20-40 LQTS patients and 10 healthy controls.

The study is ethically justified, with no extra laboratory tests or costs for participants, and written consent will be obtained from parents and capable children.

The results are expected to improve the safety of propranolol treatment in LQTS children by identifying risk factors for hypoglycemia and informing preventive strategies, such as dietary guidance, use of glucose monitoring devices during illness, or considering selective beta-blockers for high-risk patients.

DETAILED DESCRIPTION:
Frequency of Hypoglycemia in Children with Beta-Blocker Treated Long QT Syndrome

What is Long QT Syndrome (LQTS)? Long QT syndrome is a rare, inherited heart condition that can cause sudden fainting episodes and increases the risk of heart arrhythmias and sudden death. It is caused by genetic changes affecting the heart's ion channels, which control electrical activity. In Finland, about 1 in 2,000 people have LQTS.

Why Beta-Blockers? Children diagnosed with LQTS are put on beta-blocker medication (usually propranolol) as infants to prevent life-threatening arrhythmias. Beta-blockers are effective but can increase the risk of low blood sugar (hypoglycemia), especially in young children.

Why Study Hypoglycemia? Hypoglycemia is a rare but potentially serious side effect of beta-blockers. Studies show that about 3% of children with LQTS on beta-blockers experience symptomatic hypoglycemia over five years, with the highest risk in young children. The most common symptom is a hypoglycemia-triggered seizure. It is not known how often mild or symptom-free low blood sugar occurs, which could affect a child's well-being and development if repeated.

Study Goals

The study aims to answer the following questions:

* How often do children with LQTS on beta-blockers experience low blood sugar, including asymptomatic episodes?
* Can dietary advice or the use of glucose monitoring devices help prevent hypoglycemic episodes?
* Are some children with LQTS more sensitive to hypoglycemia, and do genetic factors explain these differences?
* How many children with LQTS need emergency care or hospitalization due to hypoglycemia compared to healthy children?

Who Will Participate?

* 20-40 children under 7 years of age with genetically confirmed LQTS (types 1 or 2) and on beta-blocker medication.
* 10 healthy children (siblings of LQTS patients) as controls.

Children with diabetes, other metabolic diseases, tube feeding, certain medications, dialysis, or severe acute illness are excluded from the study.

Participation is voluntary. Parents are given informed consent, and children who are able are also given their own consent. Information is provided both verbally and in writing.

Study Methods Continuous Glucose Monitoring (CGM) Each child will use a CGM device (Dexcom G7) for 10 days while the child is healthy, and again for 10 days during an infection (when risk of hypoglycemia is higher due to reduced eating). If a child has hypoglycemia and receives dietary advice, a third monitoring episode may be done.

Both LQTS patients and healthy controls undergo the same CGM.

What Happens During Monitoring? If the continous glucose monitor detects low glucose (<3.1 mmol/l), a finger-prick test is done to confirm the hypoglycemia. If low glucose level is confirmed, the child is given sugar containing food or drink. Breastfed infants receive breast milk. All measurements are recorded, and electronic data is stored on HUH secure servers.

Data is analyzed to compare average glucose levels, time spent with low or high glucose and number of finger-prick confirmed hypoglycemic episodes within the groups (healthy vs infection episode) and between groups (controls vs LQT1 and 2 patients).

Dietary Intervention Children with significant hypoglycemic episodes are referred to a dietitian. Dietitians may recommend adding slow-digesting carbohydrates (like whole grain bread) and uncooked cornstarch to the diet, especially at night or during illness, to help maintain stable glucose levels.

Genetic Analysis If some children are more sensitive to hypoglycemia, researchers will use data from the Helsinki biobank to look for genetic differences affecting insulin production and glucose metabolism.

Emergency Care Data Researchers will review records of emergency visits and hospitalizations due to hypoglycemia among LQTS patients under 16 and compare these to healthy controls.

Devices Used Dexcom G7 Glucose monitoring system

The Dexcom G7 CGM system reports continuous interstitial blood glucose concentrations every 5 minutes, does not require calibration, and involves only 1 needle stick to place the sensor. Dexcom G7 CGM system alerts for low glucose sensor readings. The manufacturer recommends that a single device may be used for up to 10 days. The Dexcom G7 system is CE-marked and FDA approved CGM system for children (age >2 years).

Risks and Benefits Risks Minor pain or discomfort from continuous glucose monitoring device placement or finger-prick tests.

Possible mild skin reactions to adhesive tape. Rare risk of infection or bleeding at the device site. For infants, continuous glucose monitoring readings may be less accurate due to thinner skin, but low readings are always confirmed with a finger-prick test.

Benefits Less painful than repeated finger-prick tests. Provides more complete data on glucose levels. If low glucose is detected, care can be adjusted to improve safety (diet changes, CGM use during illness or switching medications).

Participants receive a summary of their own glucose data if they wish.

Data Handling and Privacy Paper records are stored securely until 2041. Electronic data is stored on HUH secure servers, accessible only to the research team. CGM data is uploaded to a dedicated cloud account for the project.

Study Timeline and Funding Recruitment starts in autumn 2024 and ends by late 2026. Data collection continues until June 2027. Results will be analyzed by the end of 2027. The study is funded by the Pediatric Research Foundation (25,000 euros), with additional funding sought if needed.

Participation is free for families; no compensation is paid.

Reporting and Dissemination Results will be published in international peer-reviewed journals and shared through HUSH communications, social media, and Finnish medical publications.

A final report will be submitted to authorities within a year of study completion, including device details, methods, analysis, and critical evaluation.

Ethical Considerations The study follows ethical principles for medical research involving humans and complies with all relevant laws and guidelines. No extra laboratory tests or costs for participants. Written consent is obtained from parents and children who can write. If unexpected findings are discovered, participants are referred for proper care.

Why Is This Study Important? It will provide new information about the safety of beta-blocker treatment in children with LQTS. Identifying and preventing low blood glucose episodes can improve children's well-being and neurological development. Results may lead to better dietary advice, use of continuous glucose monitoring during illness, or changes in medication for high-risk children. The study aims to improve care and safety for children with LQTS, especially those most at risk.

ELIGIBILITY:
Inclusion Criteria:

* Study group: children under 7 years of age with genetically confirmed LQTS (types 1 or 2) and on beta-blocker medication
* Control group: healthy children (siblings of LQTS patients)

Exclusion Criteria:

-Children with diabetes, inherited diseases of inborn error of metabolism, tube feeding, gastrointestinal operations with risk for dumping, medications leading to hypoglycemia, dialysis, or any severe acute illness

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time spent in low glucose (<3.9 mmol/l) | 10 days continuous glucose monitoring
  Time spent in low glucose (<3.9 mmol/l) in GCM will be compared within the LQT patient group (during healthy episode vs during an infection)

SECONDARY OUTCOMES:
Difference in time spent in very low glucose (<3.1 mmol/l) | 10 days continuous glucose monitoring
  Time spent in very low glucose (<3.1 mmol/l) in GCM will be compared within the groups (healthy vs infection episode) and between groups (controls vs LQT patients)
Time spent in low glucose (<3.9 mmol/l) between groups | 10 days continuous glucose monitoring
  Time spent in low glucose (<3.9 mmol/l) in GCM will be compared between groups (controls vs LQT patients)
Nuber of finger prick confirmed hypoglycemic episodes | 10 days continuous glucose monitoring
  If CGM alerts for low glucose (<3.1 mmol/l), a finger-prick test is done to confirm weather it is an actual hypoglycemia or false sensor reading. Number of finger-prick confirmed hypoglycemic episodes are compared within the groups (healthy vs infection episode) and between groups (controls vs LQT patients).
Number of participants with adverse outcomes at the device site | 10 days continuous glucose monitoring
  Safety of CGM device will be evaluated by the presence of irritation, infection, cellulitis, bleeding, or other concerns at the device site.

CONTACTS AND LOCATIONS:
Overall Officials: Elina Hakonen, MD, PhD, Principal Investigator — New Children's Hospital, Helsinki University Hospital
Locations (1):
- New Children's Hospital, Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carnovale C, Gringeri M, Battini V, Mosini G, Invernizzi E, Mazhar F, Bergamaschi F, Fumagalli M, Zuccotti G, Clementi E, Radice S, Fabiano V. Beta-blocker-associated hypoglycaemia: New insights from a real-world pharmacovigilance study. Br J Clin Pharmacol. 2021 Aug;87(8):3320-3331. doi: 10.1111/bcp.14754. Epub 2021 Feb 23. PMID 33506522
- [Background] Poterucha JT, Bos JM, Cannon BC, Ackerman MJ. Frequency and severity of hypoglycemia in children with beta-blocker-treated long QT syndrome. Heart Rhythm. 2015 Aug;12(8):1815-9. doi: 10.1016/j.hrthm.2015.04.034. Epub 2015 Apr 27. PMID 25929701
- [Background] Torekov SS, Iepsen E, Christiansen M, Linneberg A, Pedersen O, Holst JJ, Kanters JK, Hansen T. KCNQ1 long QT syndrome patients have hyperinsulinemia and symptomatic hypoglycemia. Diabetes. 2014 Apr;63(4):1315-25. doi: 10.2337/db13-1454. Epub 2013 Dec 18. PMID 24357532
- [Background] Koponen M, Marjamaa A, Hiippala A, Happonen JM, Havulinna AS, Salomaa V, Lahtinen AM, Hintsa T, Viitasalo M, Toivonen L, Kontula K, Swan H. Follow-up of 316 molecularly defined pediatric long-QT syndrome patients: clinical course, treatments, and side effects. Circ Arrhythm Electrophysiol. 2015 Aug;8(4):815-23. doi: 10.1161/CIRCEP.114.002654. Epub 2015 Jun 10. PMID 26063740